CLINICAL TRIAL: NCT04869020
Title: Evaluation of the OtoBand in Subjects With Self-reported Vertigo to Reduce Severity of Vertigo in a Real-world Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otolith Labs (Industry)
Responsible Party: Principal Investigator, Didier Depireux, Chief Science Officer, Otolith Labs
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Olith10701
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Vertigo
Keywords: BPPV; Meniere's disease; Migraine associated vertigo; Labyrinthitis; Vestibular neuritis
MeSH Terms: conditions — Vertigo; Meniere Disease; Labyrinthitis; Vestibular Neuronitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant will be assigned to one of the study's two arms. Participants in Arm 1 will receive, in random order, an OtoBand or Sham Device A to use for two weeks each. Participants in Arm 2 will receive, in random order, a OtoBand or Sham Device B. The participants and researchers will be blinded to which arm of the study a participant is assigned and they will not know if the device in use is effective or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Otoband efficacy versus Sham A (Other): Participants in Arm 1 will receive, in random order, an OtoBand or Sham Device A to use for two weeks each. Sham Device A is an OtoBand in which the transducer is modified so that the vibrations do not target the vestibular system. There will be a two-day washout period between the devices. For the second two weeks, the participants will receive the alternate device (i.e., sham or effective).
  Interventions: Device: Otoband; Device: Sham A
- Otoband efficacy versus Sham B (Other): Participants in Arm 2 will receive, in random order, a OtoBand or Sham Device B. Sham Device B is an OtoBand that operates at settings found to be non-therapeutic in motion sickness studies. There will be a two-day washout period between the devices. For the second two weeks, the participants will receive the alternate device (i.e., sham, or effective).
  Interventions: Device: Otoband; Device: Sham B

INTERVENTIONS:
Device: Otoband — Participants with vertigo will wear the Otoband set at their chosen power level when experiencing symptoms.
Device: Sham A — Sham Device A is an OtoBand in which the transducer is modified so that the vibrations are not targeted at the vestibular system.
  Arms: Otoband efficacy versus Sham A
Device: Sham B — Sham Device B is an OtoBand that operates at power settings found to be nontherapeutic against vertigo associated with virtual reality.
  Arms: Otoband efficacy versus Sham B

SUMMARY:
This study seeks to gather data on the effect of a device, the OtoBand, in participants who have reported symptoms of vertigo, compared to the effect of using one of two sham devices. The study is designed to be conducted remotely using video conferencing between representatives of the manufacturer of the Otoband and participants. In order to comply with requirements for non-essential contact due to the Covid-19 pandemic there will be no person to person contact in the study.

DETAILED DESCRIPTION:
In this phase of this pilot study, a minimum of 20 participants will be enrolled, with up to 100 participants maximum. This will provide adequately powered pilot data to measure effect size for the OtoBand and sham devices and to identify different causes of vertigo for which the OtoBand has a particularly strong effect as measured by the Otolith Vertigo Assessment Tool. After inclusion/exclusion screening and informed consent is obtained, potential participants will be assessed using the Dizziness Handicap Inventory (DHI). The DHI will be completed online.

Potential participants with a DHI score in the appropriate range will be accepted into the study. These participants will be asked to schedule an online meeting to with the study coordinator. In this online enrollment meeting, the study coordinator will review the Informed Consent and confirm other information supplied by the participant online (inclusion/exclusion) and then make an affirmative decision to enroll or not enroll participants in the study.

The participants will be randomly assigned to one of the two arms of the study (OtoBand / Sham Device A or OtoBand / Sham Device B). This is a blinded study in which every participant will be evaluated, and each participant may select the stimulation that best suits him or her on both of the study devices.

Each participant will select his/her preferred stimulation level by pressing the power level button on the study device; however, they will be blinded to which device they are using. Study participants will be asked to use the devices whenever they are having a symptom of vertigo. Each participant will be asked to record his/her level of vertigo in the online Study Diary: before putting on the device, after wearing the device for 5 minutes, after removing the device.

The study devices will record the following information regarding usage: Date and time when the device is turned on/off and the power level, Date and time when the power level is changed and the new power level.

Participants will be allowed to use the device as long as they are getting benefit from the device at any power setting that they select. Participants will be asked to complete an entry in the Study Diary even on days on which they do not experience a vertigo episode.

The study coordinator will schedule six study monitoring call with each participant as close as possible to the following schedule:

Call 1: Device I: 4 days after enrollment Call 2: Device I: 9 days after enrollment Call 3: Device I: 14 days after enrollment Call 4: Device II: 17 days after enrollment Call 5: Device II: 22 days after enrollment Call 6: Device II: 27 days after enrollment

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18 to 70 years old
* Vertigo that has been present for at least 90 days
* Vertigo that is constant or predictable
* Consulted a medical doctor in the past 24 months regarding their vertigo
* Identify as having vertigo from one of the following causes:
* Benign Paroxysmal Positional Vertigo (BPPV)
* Meniere's Disease
* Vestibular Migraines
* Migraine Associated Vertigo
* Vestibular Neuritis
* Labyrinthitis
* Vertigo caused by COVID-19
* Score within appropriate range on the Dizziness Handicap Inventory
* Have a computer and access to internet for online video conferences
* PayPal, Venmo or Zelle account to receive compensation

Exclusion Criteria:

* Vertigo that first presented within the last 90 days
* Skull base surgery within the last 90 days
* Any skull implant (cochlear implant, bone conduction implant, DBS)
* Taking benzodiazepines (e.g., clonazepam, lorazepam, diazepam) for dizziness
* Vitreous detachment of the retina (floaters in the eye) in the previous 90 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
Change in vertigo severity rating while wearing the OtoBand compared to the change in vertigo severity while wearing a sham device. | Forms filled out daily over four week period by the study participant
  The primary endpoint will be the change in vertigo severity rating while wearing the OtoBand compared to the change vertigo severity while wearing the sham device during the worst, most intense episode of vertigo within each treatment period (sham versus OtoBand device).

SECONDARY OUTCOMES:
Average change in vertigo severity rating while wearing the OtoBand compared to average change in vertigo severity while wearing the sham device. | Forms filled out daily over four week period by the study participant
  This secondary outcome measure will be a statistically significant average improvement in reported vertigo when wearing the OtoBand, using the average change in reported vertigo when wearing the sham device as a reference.
Frequency of vertigo events during each period of testing (OtoBand versus sham). | Forms filled out daily over four week period by the study participant
  We will compare the number of "definite vertigo days" during the study period, comparing the OtoBand period vs the sham period.
Durability of the effect over the observation period. | Forms filled out daily over four week period by the study participant
  We will compare the mean change in reported vertigo during the first week vs the second week of use, for the period of OtoBand use and the period of sham device use. This will give an indication of whether any potential therapeutic effect of the devices remains constant over the duration of the study.
Complaints regarding usage. | Information gathered in each monitoring visits over the four week period.
  We will classify complaints expressed during monitoring visits as "discomfort", "worsening" and those related to "efficacy", and model interactions between time and number of complaints, as a function of the testing group (OtoBand versus sham).
Relationship of the bone conduction stimulation level (in dB) selected by the participant to severity of reported vertigo. | Forms filled out daily by the study participant over four week period compared to two data files captured by the devices over their two week usage.
  We will evaluate any relationship between preferred bone conduction stimulation level and severity of vertigo episodes, by modelling interactions between time and (mean) bone conduction stimulation level selected by the participant for each vertigo episode, as a function of the testing group (OtoBand versus sham).
Duration of use within each episode of vertigo and over the entire observation period. | Forms filled out daily over four week period by the study participant
  We will evaluate any change in vertigo episode duration, by modelling interactions between time (day) and duration of device use per episode, as a function of the testing group (OtoBand versus sham).
Identification of a preferred dose. | Data captured by the devices over the 14 days with each device.
  We will measure the mean preferred power level per reported condition (BPPV, vestibulopathy, Meniere, Migraine associated vertigo) over all participants.
Identification of the sham device with the smallest placebo effect. | Forms filled out daily over 2 week period by the study participant with the sham in each arm.
  We will measure any potential effectiveness of the sham devices, by comparing the mean change in vertigo score with the OtoBand and with the sham, for each of the two sham devices.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Depireux, PhD, Principal Investigator — OtolithLabs
Locations (1):
- Otolith Labs, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No